CLINICAL TRIAL: NCT04223063
Title: Exercise-based Pre-habilitation in Bladder Cancer Patients Prior to Radical Cystectomy: a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ross Mason (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Ross Mason, Assistant Professor of Urology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21485
Record Dates: First submitted 2019-12-18; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
Keywords: Bladder Cancer; Urothelial Carcinoma; Chemotherapy; Neoadjuvant; Exercise prehabilitation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants allocated to the exercise intervention will engage in a multimodal, home-based program including strength and endurance exercises. Participants will initially be seen in person and instructed to begin a moderate-intensity (i.e., 3-4 on 10-point Borg Scale) walking (or preferred aerobic exercise) program for a minimum of 30 minutes/day, 3-5 days/week and perform strength exercises at least 2 days/week.
  Interventions: Behavioral: Exercise program
- Control (No Intervention): Participants allocated to the control group will not receive any formal exercise prescription or guidance, however they will be offered the opportunity to participate in a home-based intervention pending the completion of data collection.

INTERVENTIONS:
Behavioral: Exercise program — As per the intervention arm
  Other Names: Multimodal, home-based exercise program
  Arms: Exercise Intervention

SUMMARY:
The purpose of this study is to explore the feasibility and efficacy of a 12-week, home-based exercise program in bladder cancer patients undergoing curative intent neoadjuvant chemotherapy and RC.

DETAILED DESCRIPTION:
The investigators will seek to recruit 20 patients diagnosed with muscle invasive localized urothelial carcinoma of the bladder who are scheduled to receive neo-adjuvant chemotherapy prior to RC from the Queen Elizabeth Health Sciences center in Halifax, Nova Scotia. Participants will be randomly allocated to standard of care treatment versus standard of care plus a multimodal, home-based program including strength and endurance exercises. Outcomes measured will include feasibility data, patient outcomes, and post-surgical complications.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of localized muscle invasive urothelial carcinoma of the bladder (clinical stages cT2-4a, N0-1, M0);
2. treatment plan includes the administration of cisplatin-based systemic neoadjuvant chemotherapy prior to anticipated RC (typically four, 3-week cycles of cisplatin-based chemotherapy);
3. English fluency;
4. physician approval; and
5. participant willingness to participate in a 12-week, home-based exercise intervention.

Exclusion Criteria:

1. unstable or symptomatic cardiac or pulmonary disease, musculoskeletal injury or co-morbid disease that precludes ability to exercise; and
2. significant cognitive limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life in patients with bladder cancer | 12 weeks
  Health-related quality of life during neoadjuvant chemotherapy as measured using the Functional Assessment of Cancer Therapy - Bladder scale (FACT-Bl). The 39 item FACT-B provides subscale scores of physical (7-items), functional (7-items), emotional (6-items), and social/family (7-items) well-being as well as a bladder cancer specific sub-scale. The sum of scores on subscales evaluates a participants' quality of life with higher scores denoting higher quality of life.
Fatigue | 12 weeks
  Fatigue as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-F). The FACIT-F is a 13 item scale with each item measured on a 4-point Likert scale. The total score ranges from 0 to 52. High scores represent less fatigue.
Sleep quality | 12 weeks
  Sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item tool that assesses usual sleep habits during the past month. A global sleep quality score from 0 to 21 is generated with higher scores denoting worse sleep quality

SECONDARY OUTCOMES:
Post-surgical complications | 30 days post-surgery
  Post-surgical complications will be assessed using the Clavien-Dindo grading system
Post-operative length of stay | 30 days post-surgery
  Post-operative length of stay measured as the number of days from surgery until initial discharge from hospital

OTHER OUTCOMES:
Chemotherapy completion rates | 16 weeks
  Chemotherapy completion rate measured as the percentage of patients completing four cycles of neoadjuvant chemotherapy
Post-surgical readmission rates | 90 days post-surgery
  Post-surgical readmission rates as defined by any readmission to hospital within 90 days of surgery